CLINICAL TRIAL: NCT01836679
Title: A Phase II Study of Chidamide or Placebo in Combination With Carboplatin and Paclitaxel in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Chidamide in Combination With Carboplatin and Paclitaxel in Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDM204
Record Dates: First submitted 2013-04-12; First posted 2013-04-22 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Non-small-cell Lung Cancer
Keywords: Chidamide,lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Paclitaxel; Taxes; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1.The chemotherapy cycles are repeated every 3 weeks to a maximum of 4 cycles. Patients also receive Chidamide 20mg orally twice a week until disease progression,or unacceptable toxicities,or withdrawal of consent occurred.
  Interventions: Drug: Chidamide; Drug: Paclitaxel; Drug: Carboplatin
- Arm 2 (Placebo Comparator): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1.The chemotherapy cycles are repeated every 3 weeks to a maximum of 4 cycles. Patients also receive placebo orally twice a week until disease progression,or unacceptable toxicities,or withdrawal of consent occurred.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Placebo

INTERVENTIONS:
Drug: Chidamide — Given orally
  Other Names: CS055
  Arms: Arm 1
Drug: Paclitaxel — Given IV
  Other Names: Taxol; TAX
Drug: Carboplatin — Given IV
  Other Names: CBDCA; Paraplatin
Drug: Placebo — Given orally
  Other Names: PLB
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Chidamide combined with paclitaxel and carboplatin in patients with advanced non-small-cell lung cancer.

DETAILED DESCRIPTION:
The study is to evaluate efficacy which includes the progression free survival (PFS), PFS at 6 months, objective response rate, duration of response rate, overall survival and time to progression, and safety which include adverse events, vital signs, laboratory tests, of the treatment of chidamide plus paclitaxel and carboplatin in patients with advanced non small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histology or cytology confirmed non-small-cell lung cancer,stage IIIb or IV. Newly diagnosed or relapsed after surgery but have not received systemic drug therapy.Adjuvant chemotherapy after surgery should have completed for more than one year at study entry.
* Aged 18~75 years
* Epidermal growth factor receptor (EGFR) mutation negative or EGFR status is unknown
* With at least one measurable lesion
* White blood cell count≥4×10^9/L,platelet count≥100×10^9/L and hemoglobin≥11g/L
* Life expectancy >3 months
* Eastern Cooperative Oncology Group performance status of ≤1 at study entry
* Women of childbearing age should have pregnancy test negative and would like to conduct birth control during the study
* Have signed informed consent

Exclusion Criteria:

* Patients with clinically significant corrected QT interval prolongation, or ventricular tachycardia,or auricular fibrillation, or ≥Grade 2 sino-auricular heart-block,or ≥Grade 3 atrioventricular block,or myocardial infarction within one year, or congestive heart failure,or patients with symptomatic coronary disease which need to be treated by drug
* The size of fluid area detected by cardiac ultrasonography in cavum pericardium is ≥10mm during diastolic period
* Organ transplant patients
* Patients with active bleeding or new thrombotic diseases
* Patients with body temperature >38.5℃ for more than 3 days
* Total bilirubin >1.5 fold of upper limit of normal (ULN), ALT/AST>1.5 fold of ULN or serum creatine >1.5 fold of ULN
* Patients with symptomatic brain-metastasis
* Pregnant or lactating women
* Patients with mental disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 76 weeks
  PFS is measured from the start of treatment until progression or death,whichever is first met

SECONDARY OUTCOMES:
Progression-Free Survival Rate at 6 Months (6-M-PFS) | 6 months
  6-M-PFS is defined as the percentage of participants whose disease is still progression-free at the 6th month
Object Response Rate (ORR) | Response is assessed once every 6 weeks (combination therapy period) for up to 12 weeks, and once every 8 weeks (maintenance therapy period) for up to 64 weeks
  ORR is defined as percentage of participants with Complete Response and Partial Response,assessed by the investigators according to the Response Evaluation Criteria in Solid Tumors (RECIST)
Duration of Response (DOR) | From the first date of response until the date of first documented progression, assessed up to 70 weeks
  DOR is measured from the first date when criteria for response is met until the first date when the criteria for progression is met
Overall Survival (OS) | From date of randomization until the date of death from any cause, followed for up to 76 weeks
  OS is measured from the start of treatment until death
Time To Progression (TTP) during the maintenance therapy period | From the start date of maintenance therapy until the date of first documented progression, assessed up to 64 weeks
  TTP is assessed for patients who complete the 12 weeks of combination therapy. It is measured from the start of maintenance therapy until the criteria of progression is met

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (8):
- China (8):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Hebei Provincial Tumor Hospital, Shijiazhuang, Hebei
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - The first Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai Chest Hospital Affiliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - The Second People's Hospital of Sichuan, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No